CLINICAL TRIAL: NCT06380881
Title: A Single-center, Open-label, Single-arm Phase Ib Clinical Study to Evaluate the Pharmacokinetics and Pharmacodynamic Characteristics of SHR-2017 Injection in Patients With Bone Metastases
Brief Title: PK/PD Study of SHR-2017 Injection in Patients With Bone Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-2017-102
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Patients With Bone Metastases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-2017 (Experimental)
  Interventions: Drug: SHR-2017

INTERVENTIONS:
Drug: SHR-2017 — SHR-2017

SUMMARY:
To evaluate the pharmacokinetic characteristics, pharmacodynamic characteristics, safety, tolerability and immunogenicity of SHR-2017 injection in patients with bone metastases, and to evaluate the efficacy of SHR-2017 injection in the treatment of skeletal-related event and cancer pain.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Male or female, age ≥ 18 years;
3. Solid tumors confirmed by histological or cytological examination;
4. At least 1 bone metastasis from a documented tertiary A hospital during the screening period;
5. Worst pain score NRS ≥5 points when treated with a stable analgesic regimen during the baseline assessment period;
6. Received a stable anti-tumor regimen within 28 days prior to the baseline assessment period
7. During the screening period, the physical status score of the Eastern Cooperative Oncology Group (ECOG) was 0-2 points;
8. Life expectancy judged by the investigator to be at least 6 months
9. Good organ function during the screening period (repeated testing can be confirmed if necessary);
10. Female subjects of childbearing potential with negative blood pregnancy test results within 7 days prior to the first dose of study drug and not lactating.

Exclusion Criteria:

1. Previous occurrence or concomitant osteomyelitis of the jaw or osteonecrosis of the jaw, dental disease or jaw disease that is active, requiring oral surgery, dental surgery or oral surgery wound that has not fully healed, or has planned invasive dental procedures during the study;
2. History of major joint trauma or surgery within 1 year prior to enrollment
3. Cardiac dysfunction Within 6 months before enrollment;
4. Resting tachycardia or resting bradycardia on ECG at screening；
5. Subjects who have evidence of orthostatic hypotension at screening；
6. Hepatitis B surface antigen (HBSAG), hepatitis C antibody (HCVAB), human immune defect antivirus (HIV) antibody, syphilis antibody;
7. The pain of the subjects not predominantly related to a bone metastasis;
8. The subject with neurological diseases and/or mental illness and/or cognitive dysfunction ；
9. Receipt of radiopharmaceutical treatment or radiotherapy for treatment of bone metastasis within 1 month of the treatment period, and the subject who received the radiotherapy within one month before the first research drug administration
10. Subject has a history of allergic or anaphylactic reaction to mammalian -based drugs, or allergies to supplements (calcium or vitamin D supplements), or have a history of allergens of opioids, or past history of treatment or diagnostic monoclonal antibody, Or other allergies;
11. The subject participated in the treatment of other clinical trials within one month before receiving the experimental drug (except for participating in other clinical trial screening losers);
12. In the judgment of the investigator, would make the subject inappropriate for entry into this study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
The Pharmacokinetic parameters of SHR-2017 after administration, including Cmax | First dose up to 169 days post-dose
The Pharmacokinetic parameters of SHR-2017 after administration, including Tmax | First dose up to 169 days post-dose
The Pharmacokinetic parameters of SHR-2017 after administration, including AUC0-t | First dose up to 169 days post-dose
The Pharmacokinetic parameters of SHR-2017 after administration, including AUC0-∞ | First dose up to 169 days post-dose
The Pharmacokinetic parameters of SHR-2017 after administration, including t1/2 | First dose up to 169 days post-dose
The Pharmacokinetic parameters of SHR-2017 after administration, including CL/F | First dose up to 169 days post-dose
The pharmacodynamic parameter of SHR-2017 after administration include uNTX/uCr | First dose up to 169 days post-dose
The pharmacodynamic parameter of SHR-2017 after administration include β-CTX | First dose up to 169 days post-dose
The pharmacodynamic parameter of SHR-2017 after administration include BALP [Time | First dose up to 169 days post-dose

SECONDARY OUTCOMES:
Change from baseline in worst pain/average pain at the designated bone metastasis pain site after dosing | First dose up to 169 days post-dose
  Worst pain / average pain was assessed on an 11-point numeric rating scale (NRS) ,The participant described the worst pain/average pain during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain)
Incidence of skeletal-related event | First dose up to 169 days post-dose
Average daily total opioids consumption | First dose up to 169 days post-dose]

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided